CLINICAL TRIAL: NCT00983723
Title: Clinical Proteomic Research on the Brain
Brief Title: Clinical Proteomic Research for the Brain
Acronym: "CPR Brain"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Mingming Ning, MD, Co-director, Cardio-Neurology Clinic. Director, Clinical Proteomics Research Center, Massachusetts General Hospital
Other Study IDs: 2005-P-001521; R01NS067139 (NIH); NCT00682331 (obsolete NCT alias)
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Ischemic Brain Injury; Stroke; Healthy Individual; Patent Foramen Ovale (PFO); Neurovascular Injury
Keywords: Patient Foramen Ovale; PFO; Stroke; Ischemic Brain Injury; Neurovascular Disease
MeSH Terms: conditions — Stroke; Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study of plasma and urine proteomic profiles in patients with ischemic brain injury is important to better understanding of the mechanisms by which thrombolytic agents or other therapy affects clinical outcomes. The purpose of this study is to study the proteomic profile of patients with ischemic brain injury and compare it to control subjects without ischemic brain injury, subjects with other chronic neurologic diseases or systemic vascular diseases, and pre- and post- therapy which may be associated with, or predictive of, therapeutic outcome.

The investigators hypothesize that there is a unique set of proteins expressed in serum and urine in patients with ischemic brain injury that may provide a more complete understanding of ischemic brain injury pathophysiology.

Ultimately, this study may provide information of direct relevance to the medical care of a large proportion of patients with ischemic brain injury and other neurologic diseases in the future. And proteomic proteomic profile may provide important information about the roles of specific biomarkers. Perhaps the prevention of ischemic injury related complications.

ELIGIBILITY:
Case Inclusion and Exclusion Criteria:

Inclusion Criteria:

1. Ischemic brain injury within 12 hours of symptom onset;
2. Including primary ischemic brain injury from embolism or arterial occlusion or secondary due to increased ICP after trauma, subarachnoid hemorrhage.

Exclusion Criteria:

1. Patients who are hemodynamically unstable for venipunctures;
2. Anemic patients (hemoglobin < 11);
3. Children;
4. Pregnant women.

Controls Inclusion and Exclusion Criteria:

Inclusion Criteria:

1. Healthy adults without any neurologic or systemic disease;
2. Inpatient or outpatient adults with a chronic stroke (greater than 3 months) or chronic neurologic disease such as neurodegenerative disease, movement disorder, demyelinating disease;
3. Inpatient or outpatient adults with systemic vascular disease.

Exclusion Criteria:

1. Patients who are hemodynamically unstable for venipunctures;
2. Anemic patients (hemoglobin < 11);
3. Children;
4. Pregnant women.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult with acute ischemic brain injury, adults with neurological or vascular conditions other than acute stroke and healthy adults.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2005-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome and Biomarker Outcome

CONTACTS AND LOCATIONS:
Overall Officials: MingMing Ning, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Clinical Proteomics Research Center, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Clinical Proteomics Research Center — http://www.massgeneral.org/neurology/research/researchlab.aspx?id=1318